CLINICAL TRIAL: NCT00584818
Title: A Phase 2 Dose-Finding Clinical Trial of CARDIOsphere® (PB127) in Normal Volunteers and in Patients With Known or Suspected Coronary Artery Disease
Brief Title: Dose Finding Study of PB127 Ultrasound Contrast Agent in Healthy Volunteers and Patients With Coronary Artery Disease
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Point Biomedical (Industry)
Responsible Party: Tom Ottoboni PhD/Chief Operating Officer, POINT Biomedical Corp.
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 127-013
Record Dates: First submitted 2007-12-20; First posted 2008-01-02 (Estimated); Last update posted 2008-04-25 (Estimated); Status verified 2008-04

CONDITIONS: Healthy; Coronary Artery Disease
Keywords: coronary artery disease; chest pain; healthy volunteers; SPECT; angiogram; ultrasound; echocardiogram; perfusion
MeSH Terms: conditions — Coronary Artery Disease; Chest Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: PB127 for Injectable Suspension — Stages 1 & 2 0.009 - 0.204 mg/kg continuous IV during rest and stress conditions. Infusion rate of 50 - 125 mL/hr will be adjusted for image quality and diagnostic quality. Infusion limited to 60 minutes or less.
  Stage 3 - will utilize infusion rate and dose established in Stages 1 & 2. 0.062 mg/kg continuous IV infusion at 150 mL/hr during rest and 100 mL/hr during stress conditions.
  Other Names: CARDIOsphere®

SUMMARY:
The purpose of this study is to determine the dose of PB127 for detection and/or exclusion of coronary artery disease when used with cardiac ultrasound. This study also evaluates the safety of PB127.

ELIGIBILITY:
Inclusion Criteria:

Stages 1 and 2

1. Men and women
2. Ages 18 30
3. Normal volunteers
4. No history (or suspicion) of CAD

Stage 3

1. Men and women with known or suspected CAD
2. Ages 18 years and older
3. Scheduled for or undergone clinically indicated coronary angiography within 28 days prior to or following Study Day 1

   1. Coronary angiography within 28 days prior to Study Day 1 and/or SPECT must have been non-interventional
   2. Coronary angiography images available in digital format (non cine) for transmission to core laboratory
4. Scheduled for or undergone SPECT within 28 days prior to or following Study Day 1

Exclusion Criteria:

1. Unable to provide written informed consent
2. Women who are pregnant or lactating
3. Known hypersensitivity or known contraindication to:

   1. Dipyridamole
   2. Ultrasound contrast agents (including PB127 and excipients)
   3. Blood, blood products, albumin, egg whites, or protein
4. Use of caffeine or xanthine containing products within the 24 hours prior to PB127 administration on Study Day 1 (Stages 2 and 3)
5. Previous exposure to PB127
6. Inadequate echocardiographic windows
7. Heart transplant
8. Known right to left shunt, including atrial septal defect
9. History of CABG
10. Current uncontrolled ventricular tachycardia, atrial fibrillation, atrial tachycardia, or atrial flutter
11. Pacemaker or defibrillator
12. Unstable angina grade CCS Class IV severity with ongoing symptoms and/or ongoing infusion of IV nitroglycerin
13. Second degree or greater heart block
14. Hypertension (SPB >200 and/or DBP >110 mmHg on two consecutive readings within 1 hour prior to PB127 administration)
15. Hypotension (SPB <90 mmHg on two consecutive readings within 1 hour prior to PB127 administration)
16. Severe aortic stenosis (>100 mmHg peak transvalvar gradient or <0.6 cm2 estimated valve area)
17. Pulmonary edema within the 7 days prior to Study Day 1
18. Resting oxygen saturation of less than 90%
19. Q wave MI or major surgery within the 7 days prior to Study Day 1
20. PTCA within the 28 days prior to Study Day 1
21. Chronic obstructive pulmonary disease or bronchospastic airway disease which, in the opinion of the Investigator, is significant enough to contraindicate dipyridamole
22. Known history of severe pulmonary hypertension characterized by estimated pulmonary artery systolic pressure of >50 mmHg
23. Liver disease, characterized by or including one or more of the following

    1. Elevated total bilirubin > upper limit of normal
    2. Currently elevated hepatic enzymes >3X upper limit of normal
24. Medical conditions or other circumstances that would significantly decrease the chances of obtaining reliable data or achieving the study objectives (i.e., drug dependence, psychiatric disorder, dementia, or associated illness); extenuating circumstances or medical conditions that make it unlikely that a patient can complete the clinical trial or follow up evaluations; or other reasons for expected poor compliance with the clinical investigator's instructions

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 205 (Actual)
Dates: Start 2006-11; Primary Completion 2008-03 (Actual); Study Completion 2008-03 (Actual)

PRIMARY OUTCOMES:
To identify the minimum effective dose of PB127 | 24 hours
To identify the optimal stress infusion rate of PB127 | 24 hours

SECONDARY OUTCOMES:
To assess the efficacy of PB127 MPE using the dose and stress infusion rate identified in Stages 1 and 2 | 24 hours
To evaluate the safety of PB127 | 24 hours

CONTACTS AND LOCATIONS:
Overall Officials: Alexander Ehlgen, MD, PhD, Study Director — POINT Biomedical Corp.
Locations (16):
- United States (16):
  - Long Beach VA Medical Center Cardiology Division, Long Beach, California
  - University of California San Diego Division of Cardiology, San Diego, California
  - Alfieri Cardiology, Newark, Delaware
  - University of Chicago Medical Center, Chicago, Illinois
  - Midwest Cardiology Associates, Overland Park, Kansas
  - The Center for Cardiovascular Studies Kramer and Crouse Cardiology, Shawnee Mission, Kansas
  - Androscoggin Cardiovascular Associates, Auburn, Maine
  - Cardiovascular Consultants, Kansas City, Missouri
  - St. Louis University Medical Center, St Louis, Missouri
  - The Cleveland Clinic Foundation, Cleveland, Ohio
  - Oregon Health Sciences University, Portland, Oregon
  - University of Pittsburgh Cardiovascular Institute, Pittsburgh, Pennsylvania
  - Seton Healthcare Network Brackenridge Hospital, Austin, Texas
  - Austin Heart, Austin, Texas
  - Inland Cardiology, Spokane, Washington
  - Northwest Cardiovascular Research Institute Spokane Cardiology, Spokane, Washington